CLINICAL TRIAL: NCT06242249
Title: Determining Safety and Maximum Tolerated Dose (MTD) of Anti-BCMA CAR-NK Therapy in Relapsed or Refractory Multiple Myeloma
Brief Title: Anti-BCMA CAR-NK Therapy in Relapsed or Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masoud Soleimani, Professor, Shahid Beheshti University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 74932
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma, Refractory
Keywords: CAR-NK Therapy; Anti-BCMA
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relapsed or Refractory Multiple Myeloma (Experimental)
  Interventions: Biological: Anti-BCMA CAR-NK

INTERVENTIONS:
Biological: Anti-BCMA CAR-NK — Ten eligible patients with relapsed refractory multiple myeloma will be enrolled based on inclusion criteria and informed consent. After conditioning with Fludarabine and Cyclophosphamide, patients will receive a single infusion of BCMA CAR NK cells with close monitoring using one of the following dose levels:
  * Dose Level 1: 1×10^7/Kg
  * Dose Level 2: 5×10^7/Kg
  * Dose Level 3: 1×10^8/Kg Safety Assessment: Adverse events will be recorded and graded. Laboratory parameters and cytokine release syndrome (CRS) markers will be closely monitored. Efficacy Evaluation: Response assessments will follow IMWG guidelines, including complete response (CR), partial response (PR), stable disease (SD), and progressive disease.

SUMMARY:
Immunotherapy has shown promise in the treatment of hematological malignancies, including multiple myeloma. One approach is CAR-NK cell therapy, which involves genetically modifying natural killer (NK) cells to target specific cancer antigens. While CAR-NK therapy offers advantages over CAR-T therapy, such as reduced immune system reactions and lower production time and cost, challenges remain in terms of antitumor efficacy and the tumor microenvironment. Preclinical and early clinical studies have targeted various antigens, including BCMA, with CAR-NK cells in multiple myeloma. To further investigate the potential of BCMA-targeted CAR-NK cell therapy, this study aims to evaluate its safety and determine the maximum tolerated dose (MTD) in patients who have not responded to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years with expected survival > 3 months.
2. Confirmed diagnosis of active multiple myeloma with detectable BCMA expression in malignant cells.
3. Relapsed or refractory disease with at least 2 prior lines of treatment, including a proteasome inhibitor and immunomodulator, without achieving significant efficacy.
4. Measurable disease at screening according to IMWG criteria, as defined by any of the following: Serum monoclonal paraprotein (M-protein) level ≥1.0 g/dL or urine M-protein level being as defined； or light chain MM without measurable disease in the serum or the urine； serum immunoglobulin free light chain disease dL and abnormal serum immunoglobulin kappa/lambda free light chain ratio
5. ECOG performance status of 0-1.
6. Acceptable cardiac, liver, and kidney function.
7. Signed written informed consent.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Uncontrolled active infection, HIV infection, or positive syphilis serology reaction.
3. Active hepatitis B or hepatitis C infection.
4. Recent or current use of glucocorticoids or other immunosuppressors.
5. Severe cardiac, liver, renal insufficiency, diabetes, or other diseases.
6. Participation in other clinical research in the past three months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLTs) | 4 weeks
  Incidence of dose-limiting toxicity (DLTs) within 4 weeks after infusion, characterized by >= Grade 3 signs/symptoms according to CTCAE v4.03, to assess safety and tolerability.
Assessment of Maximum Tolerated Dose (MTD) | 4 weeks
Overall Remission Rate (ORR) | 8 weeks
  Overall Remission Rate (ORR) two months after infusion, assessed using International Myeloma Working Group (IMWG) criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 48 weeks
  Progression-free survival (PFS) for up to 12 months, assessed using IMWG criteria.
Duration of Response (DOR) | 48 weeks
  Duration of Response (DOR) for up to 12 months, assessed using IMWG criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shariati Hospital, Tehran, Iran